CLINICAL TRIAL: NCT00002489
Title: PROTOCOL FOR THE TREATMENT OF MALIGNANT NON-TESTICULAR GERM CELL TUMORS
Brief Title: Combination Chemotherapy in Treating Children With Non-testicular Malignant Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 91-119; CDR0000077384 (Registry Identifier: PDQ (Physician Data Query)); NCI-V92-0021
Record Dates: First submitted 1999-11-01; First posted 2004-08-30 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Extragonadal Germ Cell Tumor; Ovarian Cancer
Keywords: stage II ovarian germ cell tumor; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; ovarian teratoma; extragonadal germ cell tumor
MeSH Terms: conditions — Ovarian Neoplasms; Teratoma, Ovarian | interventions — Dactinomycin; Filgrastim; Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Leucovorin; Methotrexate; Vincristine

INTERVENTIONS:
Biological: dactinomycin
Biological: filgrastim
Drug: carboplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: leucovorin calcium
Drug: methotrexate
Drug: vincristine sulfate
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating children who have non-testicular malignant germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of cyclophosphamide, carboplatin, and etoposide in patients with non-testicular malignant germ cell tumors. II. Improve the quality of life of these patients by shortening the length of treatment and the extent of initial surgical resection. III. Determine whether histologic subtypes have prognostic significance. IV. Determine the efficacy of short term chemotherapy in this patient population. V. Determine the role of second look surgery in predicting curability of non testicular germ cell tumors. VI. Determine the role of dose intensification of cyclophosphamide and the introduction of doxorubicin, methotrexate, and dactinomycin for those patients with partial response, no response, or progressive disease at the time of second look surgery.

OUTLINE: Patients undergo treatment on Regimen A consisting of surgical resection of tumor as appropriate for disease followed by chemotherapy with cyclophosphamide IV over 20 minutes on day 1, carboplatin IV on day 2, and etoposide IV on days 2-4. Patients receive filgrastim (G-CSF) subcutaneously (SQ) daily beginning 24-48 hours following the last dose of etoposide and continuing for 14 days or until blood counts recover (a total of 28 days). Chemotherapy repeats every 3 weeks for 4 courses in the absence of disease progression. At week 11, patients undergo second look surgery to evaluate response and resect any residual disease. Patients with no residual disease receive no further therapy. Patients with good partial response or no response receive salvage chemotherapy on Regimen B. Patients receive salvage chemotherapy on Regimen B consisting of dactinomycin IV on days 1-3, doxorubicin IV and vincristine IV continuously on days 1-3, and G-CSF SQ daily beginning 24-48 hours following last dose of vincristine and continuing for 14 days or until blood counts recover. At week 3, patients receive cyclophosphamide IV on days 1-2, vincristine IV and doxorubicin IV continuously on days 1-3 and G-CSF as previously given in Regimen B. At week 6, patients receive methotrexate IV on day 1 and leucovorin calcium orally or IV every 6 hours for 3 days, beginning 16 hours after the completion of methotrexate. At week 8, salvage chemotherapy repeats for an additional course. Patients achieving complete response following salvage chemotherapy receive no further therapy. Patients with no response are removed from study.

PROJECTED ACCRUAL: A maximum of 25 patients will be accrued for this study over 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Malignant germ cell tumors of the following stages and primary sites: Stage II/III/IV ovarian tumors Grade II/III immature glial teratomas Stage II/III/IV mediastinal tumors Stage II/III/IV presacral tumors and tumors of other primary sites No intracranial or testicular primary sites

PATIENT CHARACTERISTICS: Age: Child Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: Not specified

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1991-10; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norma Wollner, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States